CLINICAL TRIAL: NCT05242471
Title: A Phase 2b Randomized, Double-blind, Active-and Placebo-controlled, Parallel-group, Multicenter Study to Evaluate the Efficacy and Safety of Induction and Maintenance Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Combination Therapy With Guselkumab and Golimumab in Participants With Moderately to Severely Active Crohn's Disease
Acronym: DUET-CD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109178; 78934804CRD2001 (Other: Janssen Research & Development, LLC); 2021-003314-39 (EudraCT Number); 2023-504741-32-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-02-15; First posted 2022-02-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab; golimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo subcutaneously (SC). All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Drug: Placebo
- Group 2: Guselkumab (Experimental): Participants will receive guselkumab dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: Guselkumab
- Group 3: Golimumab (Experimental): Participants will receive golimumab dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: Golimumab
- Group 4: JNJ-78934804 (High-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 1 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804
- Group 5: JNJ-78934804 (Mid-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 2 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804
- Group 6: JNJ-78934804 (Low-dose) (Experimental): Participants will receive JNJ-78934804 dose regimen 3 SC. All participants who meet inadequate response criteria will be escalated to an active treatment. Participants who are eligible and willing to continue the study intervention that they are receiving at Week 44 may enter the long-term extension.
  Interventions: Biological: JNJ-78934804

INTERVENTIONS:
Biological: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Arms: Group 2: Guselkumab
Biological: Golimumab — Golimumab will be administered as subcutaneous injection.
  Arms: Group 3: Golimumab
Biological: JNJ-78934804 — JNJ-78934804 will be administered subcutaneously as per defined regimen.
  Arms: Group 4: JNJ-78934804 (High-dose); Group 5: JNJ-78934804 (Mid-dose); Group 6: JNJ-78934804 (Low-dose)
Drug: Placebo — Placebo will be administered as subcutaneous injection.
  Arms: Group 1: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-78934804 at Week 48 compared to guselkumab and golimumab.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Crohn's disease (CD) for at least 3 months prior to baseline
* Confirmed diagnosis of moderate to severe CD as assessed by Crohn'

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 703 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2029-11-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Clinical Remission at Week 48 | Week 48
  Percentage of participants with clinical remission at Week 48 will be reported. Clinical remission is based on the Crohn's Disease Activity Index (CDAI).
Percentage of Participants with Endoscopic Response at Week 48 | Week 48
  Percentage of participants with endoscopic response at Week 48 will be reported. Endoscopic response is based on change from baseline in the simple endoscopic score for Crohn's disease (SES-CD), as assessed by central endoscopy reading.

SECONDARY OUTCOMES:
Percentage of Participants with Patient-reported Outcomes (PRO)-2 Remission at Week 48 | Week 48
  Percentage of participants with PRO-2 remission at Week 48 will be reported. PRO-2 remission is based on the average daily abdominal pain (AP) and stool frequency (SF) scores.
Percentage of Participants with Endoscopic Remission at Week 48 | Week 48
  Percentage of participants with endoscopic remission at Week 48 will be reported. Endoscopic remission is based on the SES-CD, as assessed by central endoscopy reading.
Percentage of Participants with Corticosteroid-Free Clinical Remission at Week 48 | Week 48
  Percentage of participants with corticosteroid-free (60-day) clinical remission at Week 48 will be reported.
Secondary Comparison: Percentage of Participants with Clinical Remission at Week 48 | Week 48
  Percentage of participants with clinical remission at Week 48 will be reported. Clinical remission is based on the Crohn's Disease Activity Index (CDAI).
Secondary Comparison: Percentage of Participants with Endoscopic Response at Week 48 | Week 48
  Percentage of participants with endoscopic response at Week 48 will be reported. Endoscopic response is based on change from baseline in the SES-CD, as assessed by central endoscopy reading.
Percentage of Participants with Adverse Events (AEs) | Up to Week 48
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Percentage of Participants with Serious Adverse Events (SAEs) | Up to Week 48
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.
Clinical Laboratory Parameters Over Time | Up to Week 48
  Clinical laboratory parameters over time will be reported.
Vital Sign Parameters Over Time | Up to Week 48
  Vital sign parameters over time will be reported.
Suicidal Ideation Assessment Using Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to Week 48
  The C-SSRS scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Worsening of suicidal ideation is defined as an increase in severity of suicidal ideation from baseline.
Serum Concentrations of Guselkumab Over Time | Up to Week 48
  Serum concentrations of guselkumab over time will be reported. Serum samples will be analyzed to determine concentrations of guselkumab using a validated, specific, and sensitive method.
Serum Concentrations of Golimumab Over Time | Up to Week 48
  Serum concentrations of golimumab over time will be reported. Serum samples will be analyzed to determine concentrations of golimumab using a validated, specific, and sensitive method.
Percentage of Participants with Antibodies to Guselkumab | Up to Week 48
  Percentage of participants with antibodies to guselkumab will be reported.
Titers of Antibodies to Guselkumab | Up to Week 48
  Titers of antibodies to guselkumab will be reported.
Percentage of Participants with Antibodies to Golimumab | Up to Week 48
  Percentage of participants with antibodies to golimumab will be reported.
Titers of Antibodies to Golimumab | Up to Week 48
  Titers of antibodies to golimumab will be reported.
Percentage of Participants with Neutralizing Antibodies to Guselkumab. | Up to Week 48
  Percentage of participants with neutralizing antibodies to guselkumab will be reported.
Percentage of Participants with Neutralizing Antibodies to Golimumab | Up to Week 48
  Percentage of participants with neutralizing antibodies to golimumab will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (454):
- United States (90):
  - University of Alabama Liver Center, Birmingham, Alabama
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Moore Clinical Trials, LLC, Little Rock, Arkansas
  - Om Research LLC, Apple Valley, California
  - Valley Gastroenterology Medical Group, Arcadia, California
  - Southern California Research Center, Coronado, California
  - Desert Gastroenterology Associates, Lancaster, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - UCLA, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California
  - UCI Irvine Medical Center, Orange, California
  - Medical Associates Research Group, Inc., San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Pioneer Research Solutions Inc., Coconut Creek, Florida
  - Homestead Associates in Research Inc, Homestead, Florida
  - Osceola Mental Health D/B/A Park Place Behavioral Health Care, Kissimmee, Florida
  - Florida Research Center Inc., Lakewood Rch, Florida
  - University of Miami Hospital, Miami, Florida
  - Gastroenterology Group Of Naples, Naples, Florida
  - Omega Research Consultants, Orlando, Florida
  - Synergy Clinical Research, St. Petersburg, Florida
  - GCP Clinical Research, Tampa, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University of Mississippi Medical Center, Atlanta, Georgia
  - Gastroenterolgy Associates of Central GA, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, Marietta, Georgia
  - Northwestern University, Chicago, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - Gastroenterology of Southern Indiana, New Albany, Indiana
  - Cotton O'Neil Digestive Health Center, Topeka, Kansas
  - Ascension via Christi Research, Wichita, Kansas
  - Univ. of KS School of Med, Wichita, Kansas
  - Tri-State Gastroenterology Assoc, Crestview Hills, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Lahey Hospital & Medical Center, Boston, Massachusetts
  - Brigham And Women's Hospital, Chestnut Hill, Massachusetts
  - FC Research, LLC, South Dartmouth, Massachusetts
  - Detroit Clinical Research Center, Livonia, Michigan
  - Huron Gastroenterology Associates Center for Digestive Care, Ypsilanti, Michigan
  - Gastrointestinal Associates LLP, Flowood, Mississippi
  - Washington University, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Care Access Las Vegas, Las Vegas, Nevada
  - Dartmouth Hitchcock, Lebanon, New Hampshire
  - Northwell Health, Great Neck, New York
  - A1 Clinical Research, Jackson Heights, New York
  - Weill Cornell Medical College, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Mohawk Valley Endoscopy Center, Utica, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Tryon Medical Group, Charlotte, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Northshore Gastroenterology Research, LLC, Westlake, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Susquehanna Gastroenterology Associates, Harrisburg, Pennsylvania
  - University of Pennsylvania - Perelman School of Medicine, Philadelphia, Pennsylvania
  - Frontier Clinical Research, Smithfield, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Digestive Disease Associates, Rock Hill, South Carolina
  - Saint Francis Hospital, Germantown, Tennessee
  - Galen Medical Group, Hixson, Tennessee
  - Etsu Quillen College Of Medicine, Johnson City, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Amel Med LLC Research, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Accurate Clinical Research, Houston, Texas
  - Gastroenterology Clinic Of San Antonio P A, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Digestive Health Specialists, Tyler, Texas
  - Care Access Research, Ogden, Ogden, Utah
  - Care Access Research- Salt Lake City, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Hunter Holmes McGuire Veterans Affairs Medical Center, Richmond, Virginia
  - Washington Gastroenterology, PLLC, Bellevue, Washington
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Digestive Disease Center, Seattle, Washington
  - Digestive Health Specialists, Tacoma, Washington
  - Marshall Health Clinical Research Center, Huntington, West Virginia
- Australia (10):
  - The Queen Elizabeth Hospital, Adelaide
  - Box Hill Hospital, Box Hill
  - Monash Health, Monash Medical Centre, Clayton
  - Western Health, Footscray
  - St Vincent's hospital, Melbourne
  - Royal Prince Alfred Hospital, Newtown
  - Royal Adelaide Hospital, North Terrace
  - Royal Melbourne Hospital, Parkville
  - Nepean Hospital, Penrith
  - Mater Hospital Brisbane Inflammatory Bowel Diseases, South Brisbane
- Austria (3):
  - Landeskrankenhaus Salzburg, Universitätsklinik f. Innere Medizin III, Salzburg
  - Akh Wien, Vienna
  - Klinikum Wels Grieskirchen, Wels
- Belgium (10):
  - GZA Ziekenhuizen, Antwerp
  - Algemeen Ziekenhuis Sint-Jan, Bruges
  - Cliniques Universitaires Saint Luc, Brussels
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
  - CHC MontLegia, Liège
  - CHU de Liege, Liège
  - Az Sint-Maarten, Mechelen
  - Algemeen Ziekenhuis Delta, Roeselare
  - Vitaz, Sint-Niklaas
- Brazil (23):
  - Hospital Das Clinicas Da Ufmg, Belo Horizonte - MG
  - Fundacao para o Desenvolvimento Medico Hospitalar (UNESP Botucatu), Botucatu
  - Impar Servicos Hospitalares S/A - Hospital Brasilia, Brasília
  - Chronos Clinica Medica Ltda, Brasília
  - Centro Digestivo de Curitiba - Instituto de Pesquisa Clínica, Curitiba
  - Centro de Estudos Clínicos do Interior Paulista - CECIP, Jaú
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Associacao Hospitalar Moinhos de Vento, Porto Alegre
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - NPCRS Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Universidade Federal do Rio de Janeiro - Faculdade de Medicina, Rio de Janeiro
  - Pesquisare Saude, Santo André
  - Irmandade da Santa Casa da Misericórdia de Santos, Santos
  - Kaiser Hospta, São José do Rio Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo
  - Hospital Nove de Julho, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual IAMSPE, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Hepatogastro, São Paulo
  - BR Trials, São Paulo
- Bulgaria (2):
  - UMHAT 'Aleksandrovska' EAD, Sofia
  - MHAT Tzaritza Joanna, Sofia
- Canada (22):
  - Foothills Hospital, Calgary, Alberta
  - Gastroenterology and Internal Medicine Research Institute (GIRI), Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Covenant Health/Grey Nuns hospital, Edmonton, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - The Gordon & Leslie Diamond Health Care Center, Vancouver, British Columbia
  - GIRI Gastrointestinal Research Institute, Vancouver, British Columbia
  - The Medical Arts Health Research Group, Vancouver, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - Winnipeg Health Sciences Centre, Winnipeg, Manitoba
  - Viable Clinical Research, Dartmouth, Nova Scotia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Barrie GI Associates, Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - Toronto Immune and Digestive Health Institute Inc, Toronto, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
  - McGill University - Health Centre - Montreal General Hospital, Montreal, Quebec
  - St. Jerome Medical Research, Saint-Jérôme, Quebec
  - CMIIM, Centre médical L'Enjeu, Ville Mont-Royal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
  - Viable Clinical Research, Bridgewater
  - Hopital Chicoutimi, Saguenay
- China (24):
  - China Japan Friendship Hospital, Beijing
  - The second Xiangya Hospital of Central South University, Changsha
  - Changzhou No 2 Peoples Hospital, Changzhou
  - West China Hospital Sichuan University, Chengdu
  - Chongqing Medical University, Chongqing
  - The First People's Hospital of Foshan, Foshan
  - Sun Yat-sen University - The Sixth Affiliated Hospital Guangdong Gastrointestinal Hospital, Guangzhou
  - Guangzhou First Municipal People's Hospital, Guangzhou
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Jinhua municipal central hospital, Jinhua
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Nanjing Drum Tower Hospital, Nanjing
  - Shanghai East Hospital, Shanghai
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
  - The Central Hospital of Wuhan, Wuhan
  - Wuhan Union Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - Wuxi People s Hospital, Wuxi
  - Zhongshan Hospital, Xiamen University, Xiamen
  - Yangzhou First People's Hospital, Yangzhou
  - ZhuZhou Central Hospital, Zhuzhou
- Croatia (3):
  - Opca bolnica Bjelovar, Bjelovar
  - University Hospital Center Split, Split
  - University Hospital Dubrava, Zagreb
- Czechia (3):
  - Vojenska nemocnice Brno, Brno
  - ISCARE a.s., Prague
  - Detska klinika Masarykovy nemocnice v Usti nad Labem, Ústí nad Labem
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg Og Frederiksberg Hospital, Copenhagen
  - Herlev Hospital, University of Copenhagen, Herlev
  - Odense Universitetshospital, Odense
  - Silkeborg Hospital, Silkeborg
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn
  - Tallinn Children's Hospital, Tallinn
  - Tartu University Hospital, Tartu
- France (15):
  - CHU Amiens - Hopital Sud, Amiens
  - CHRU De Besancon, Besançon
  - Centre Hospitalier Universitaire(CHU) - Hopital Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - Hopital Nord Marseille, Marseille
  - CHU de Nantes hotel Dieu, Nantes
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - CHU de Nice Hopital de l Archet, Nice
  - Hopital Saint Louis - Service de Gastro-Entérologie, 1 Avenue Claude Vellefaux, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHRU Hopital de Pontchaillou, Rennes
  - Hôpital Yves Le Foll, Saint-Brieuc
  - Centre hospitalier universitaire de St Etienne, Saint-Etienne
  - CHU Rangueil, Toulouse
  - CHRU Nancy Brabois, Vandœuvre-lès-Nancy
- Germany (42):
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
  - Praxis Fur Gastroenteroligie, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Krankenhaus Waldfriede Mitte, Berlin
  - Evangelisches Krankenhaus Kalk, Cologne
  - Medizinisches Versorgungszentrum (MVZ) Dachau, Dachau
  - University Hospital Dresden, Dresden
  - MVZ Sanaklinikum Duisburg, Duisburg
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum Essen, Essen
  - JWG-University Hospital, Frankfurt
  - Agaplesion Frankfurter Diakonie Kliniken GmbH, Markus Krankenhaus, Frankfurt am Main
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Fulda - Tumorklinik - Germany, Fulda
  - Curiositas ad Sanum Studien und Beratungs GmBH, Haag
  - Martin-Luther-Universitaet Halle-Wittenberg - Universitaetsk, Halle
  - BSF Studiengesellschaft, Halle
  - CTC North GmbH & Co. KG, Am Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Gastroenterology Outpatient Clinic Prof. Ehehalt/Dr. Hemstäd, Heidelberg
  - University Hospital Heidelberg, Heidelberg
  - Universitatsklinikum Jena, Jena
  - Praxisgemeinschaft Jerichow, Jerichow
  - Gastroenterologische Spezialpraxis - Berlin-Karlshorst, Karlshorst
  - Gastroenterologie Opernstrasse, Kassel
  - Universitatsklinikum Schleswig Holstein Kiel, Kiel
  - Eugastro GmbH, Leipzig
  - Staedtisches Klinikum Lueneburg, Lüneburg
  - Medizinische Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Gastroenterologische Gemeinschaftspraxis Minden, Minden
  - Klinikum der Universitaet Muenchen, Munich
  - Universitatsklinikum Munster, Münster
  - MVZ Portal 10, Münster
  - Tumorzentrum Nordthüringen Medizinisches Versorgungszentrum, Nordhausen
  - Medius Klinik Nurtingen, Nürtingen
  - Siloah St Trudpert Klinikum, Pforzheim
  - Universitaetsklinikum Regensburg, Regensburg
  - Universitaetsmedizin Rostock, Rostock
  - Zentrum für Gastroenterologie Saar MVZ GmbH, Saarbrücken
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Universitatsklinikum Wurzburg, Würzburg
- Greece (3):
  - General Hospital of Athens 'Ippokrateion', Athens
  - Sotiria General State Hospital of Chest Diseases, Athens
  - Hippokration Hospital, Thessaloniki
- Hungary (6):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Semmelweis Egyetem, Budapest
  - Semmelweis Egyetem I.Belgyogyaszati Klinika, Budapest
  - Bugat Pal Korhaz, Gyöngyös
  - Szegedi Tudomanyegyetem, Szeged
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- India (12):
  - ICON Hospital Orchid Medi services and Research Private Limited, Ahmedabad
  - M S Ramaiah Medical College and Hospital, Bengaluru
  - Siksha O Anusandhan University - Institute of Medical Scienc, Bhubaneswar
  - Srm Institutes For Medical Science (Sims), Chennai
  - Fortis Memorial Research Institute, Gurugram
  - Asian Institute Of Gastroenterology, Hyderabad
  - Yashoda Super Speciality Hospitals, Hyderabad
  - P D Hinduja National Hospital and Medical Research Center, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Yashoda Super Speciality Hospitals, Secunderabad
  - Surat Institute of Digestive Sciences Hospitals, Surat
  - Gujarat Gastro and Vascular Hospital, Surat
- Israel (10):
  - Haemek Medical Center - Afula, Afula
  - Bnai Zion Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah Hebrew University Medical Center, Jerusalem
  - Rabin Med Ctr Beilinson Hosp, Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Assaf Harofeh Medical Center, Tzrifin
- Italy (12):
  - Università degli Studi di Bari, Bari
  - A.O. Per L' Emergenza Cannizzaro - U.O. Chirurgia Generale, Catania
  - AOU Policlinico G.Martino, Messina
  - Ospedale San Raffaele, Milan
  - Ospedale Specializzato in Gastroenterologia Saverio de Bellis, Monopoli
  - Azienda Ospedaliero Universitaria di Cagliari - Policlinico Duilio Casula di Monserrato, Monserrato
  - Azienda Ospedaliera San Gerardo, Monza
  - Ospedale Classificato Equiparato Sacro Cuore Don Calabria di Negrar, Negrar ( Ve)
  - Ospedale Villa Sofia-Cervello, Palermo
  - Catholic University of Sacred Hearth, Roma
  - IRCCS Humanitas Rozzano-IBD Center Malattie Infiammatorie Croniche Intestinali, Rozzano
  - Ospedale Molinette, AO Città della Salute e della Scienza di, Torino
- Japan (53):
  - Asahikawa Medical University Hospital, Asahikawa
  - Tokyo Medical and Dental University Hospital, Bunkyō City
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Hospital of the University of Occupational and Enviromental Health, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Tokai University Hachioji Hospital, Hachiōji
  - Hamamatsu University Hospital, Hamamatsu
  - National Hospital Organization Hirosaki General Medical Center, Hirosaki
  - Hirosaki University Hospital, Hirosaki
  - Hitachi General Hospital, Hitachi
  - Hyogo Medical University Hospital, Hyōgo
  - Kagoshima University Hospital, Kagoshima
  - Kagoshima IBD Gastroenterology Clinic, Kagoshima
  - Ofuna Chuo Hospital, Kamakura
  - Kanazawa University Hospital, Kanazawa
  - Tsujinaka Hospital Kashiwanoha, Kashiwa
  - Saitama Medical University Saitama Medical Center, Kawagoe
  - Kyushu Rosai Hospital, Kitakyushu
  - Kobe University Hospital, Kobe
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyorin University Hospital, Mitaka
  - Iwate Medical University Hospital, Morioka
  - Nagaoka Red Cross Hospital, Nagaoka
  - Nagasaki University Hospital, Nagasaki
  - Nagoya University Hospital, Nagoya
  - Niigata University Medical And Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Kinshukai Infusion Clinic, Osaka
  - Osaka City University Hospital, Osaka
  - Japan Community Health Care Organization Osaka Hospital, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saga University Hospital, Saga
  - Tokitokai Tokito Clinic Coloproctology Center, Saitama
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Tokushukai Hospital, Sapporo
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo
  - Sapporo Medical University Hospital, Sapporo
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga-gun
  - Jichi Medical University Hospital, Shimotsuke
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku Ku
  - Tokyo Women's Medical University Hospital, Shinjuku-Ku
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - Takamatsu Red Cross Hospital, Takamatsu
  - The Jikei University Hospital, Tokyo
  - Kitasato University Kitasato Institute Hospital, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Ieda Hospital, Toyota
  - Mie University Hospital, Tsu
  - Yokohama City University Medical Center, Yokohama
- Jordan (4):
  - Jordan University Hospital, Amman
  - Abdali Hospital, Amman
  - Irbid Specialty Hospital, Irbid
  - King Abdullah University Hospital, Irbid
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Ampang, Ampang
  - Hospital Pulau Pinang, George Town
  - University Malaya Medical Centre, Kuala Lumpur
- Netherlands (6):
  - Academisch Medisch Centrum Universiteit van Amsterdam, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Leiden University Medical Center, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Erasmus MC, Rotterdam
  - UMC Utrecht, Utrecht
- New Zealand (3):
  - Dunedin Hospital, Dunedin
  - Hutt Hospital, Lower Hutt
  - Wellington Hospital, Wellington
- Norway (5):
  - Alesund sjukehus, Ålesund
  - Vestre Viken HF Baerum Sykehus, Gjettum
  - Akershus Universitetssykehus, Lørenskog
  - Oslo University Hospital HF Ulleval sykehus, Oslo
  - Universitetssykehuset Nord-Norge HF, Tromsø
- Poland (21):
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Centrum Medyczne Promed, Krakow
  - AmiCare Centrum Medyczne, Lodz
  - Gastromed ZOZ, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Synexus Polska Sp z o o, Poznan
  - Twoja Przychodnia, Poznan
  - Centrum Medyczne Medyk, Rzeszów
  - Endoskopia Sp z o.o., Sopot
  - Sonomed Sp. z o.o., Szczecin
  - GASTROMED Sp. z o.o., Torun
  - Centrum Zdrowia Matki Dziecka i Mlodziezy, Warsaw
  - Centralny Szpital Kliniczny Mswia, Warsaw
  - Reumatika-Centrum Reumatologii, NZOZ, Warsaw
  - NZOZ Vivamed, Warsaw
  - Bodyclinic Sp. z o.o. sp. k, Warsaw
  - Melita Medical Sp. z o.o., Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
  - Centrum Diagnostyczno - Lecznicze Barska sp. z o.o. Szpital Specjalistyczny Barska, Włocławek
  - ETG Zamosc, Zamość
- Portugal (4):
  - Centro Hospitalar Lisboa Norte EPE Hosp. Santa Maria, Lisbon
  - Hospital de Portimao-Centro Hospitalar do Barlavento Algarvio, Portimão
  - Centro Hospitalar Vila Nova de Gaia, Porto
  - Centro Hospitalar de Entre o Douro e Vouga, E.P.E, Santa Maria da Feira
- Singapore (4):
  - Singapore General Hospital, Singapore
  - KL Ling Gastroenterology and Liver Clinic, Singapore
  - Gi Associates Gastroenterology, Singapore
  - Tan Tock Seng Hospital, Singapore
- Slovenia (2):
  - Splosna bolnisnica Celje, Celje
  - Univerzitetni klinicni center Ljubljana, Ljubljana
- South Africa (6):
  - Worthwhile Clinical Trials Lakeview Hospital, Benoni
  - Mediclinic Panorama, Cape Town
  - Inspired GI Care, Cape Town
  - Clinical Research Centre University of Cape Town, Cape Town
  - Groote Schur Hospital, Cape Town
  - Hillcrest private, Durban
- South Korea (16):
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Dongguk University Ilsan Hospital, Goyang-si
  - Chosun university hospital, Gwangju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea Seoul St.Mary's Hospital, Seoul
  - Kyung Hee University Hospital, Seoul
  - The Catholic University of Korea, Suwon
  - Ajou University Hospital, Suwon
- Spain (6):
  - Hosp. Univ. La Paz, Madrid
  - Hosp. de Navarra, Pamplona
  - Hosp. Montecelo, Pontevedra
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Univ. de Torrejon, Torrejón de Ardoz
- Sweden (3):
  - Universitetssjukhuset Orebro, Örebro
  - Karolinska University Hospital, Solna
  - Ersta sjukhus, Stockholm
- Switzerland (5):
  - Universitatsspital Basel, Basel
  - Inselspital Universitatsspital Bern, Bern
  - Gastroenterologische Praxis Balsiger und Seibold, Bern
  - Kantonsspital St Gallen, Sankt Gallen
  - UniversitaetsSpital Zuerich, Zurich
- Taiwan (4):
  - Chang-Hua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (10):
  - Royal Victoria Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Velocity Clinical Research, High Wycombe
  - Whipps Cross University Hospital, London
  - St Georges Healthcare NHS Trust, London
  - John Radcliffe Hospital, Oxford
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency